CLINICAL TRIAL: NCT02367729
Title: Efficacy of Auricular Neurostimulation for Adolescents With Pain-Associated Functional Gastrointestinal Disorders
Brief Title: Efficacy of Ear Neurostimulation for Adolescents With Functional Abdominal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: American Neurogastroenterology and Motility Society (Other)
Responsible Party: Principal Investigator, Katja Kovacic, MD, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KovacicK
Record Dates: First submitted 2015-02-01; First posted 2015-02-20 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Functional Disorder of Intestine; Nausea Persistent
MeSH Terms: interventions — Implantable Neurostimulators

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurostimulator (Experimental): Auricular neurostimulator treatment x 5 days each week for 4 consecutive weeks
  Interventions: Device: Neurostimulator
- Sham Neurostimulator (Sham Comparator): Inactive auricular neurostimulator treatment x 5 days each week for 4 consecutive weeks
  Interventions: Device: Sham

INTERVENTIONS:
Device: Neurostimulator — Non-invasive, battery operated neurostimulator of the external ear worn for 5 days each week x 4 weeks.
  Arms: Neurostimulator
Device: Sham — Inactive neurostimulator device pre-programmed to be inactive. To be worn for 5 days each week x 4 weeks.
  Arms: Sham Neurostimulator

SUMMARY:
This study evaluates the effectiveness of a neurostimulator applied to the outer ear for adolescents with functional gastrointestinal disorders. The neurostimulator provides nerve stimulation to a branch of the vagus nerve which is thought to be involved in transmission of pain signals. Half of the study subjects will receive an active nerve stimulator while the other half will receive an inactive one.

DETAILED DESCRIPTION:
The vagus nerve innervates the gastrointestinal tract and influences the autonomic nervous system. It is thought to carry signals of discomfort and nausea to the brain where it is interpreted. The autonomic nervous system may be in imbalance in patients with functional gastrointestinal disorders. By stimulating a branch of the vagus nerve in the outer ear, this study aims to improve symptoms and quality of life in adolescents with functional abdominal pain with or without nausea.

Subjects will be randomized into two groups: 1) neurostimulation versus 2) sham. They will receive either an active or non-active (sham group) device for 5 days each week x 4 weeks total. Pain, nausea, anxiety, quality of life, potential side effects and overall symptom improvement will be monitored weekly for the entire study as well as after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with a major complaint of abdominal pain (minimum 3/10 in severity) with or without nausea (minimum 3/10 in severity) of unclear etiology, who are English-speaking and willing to participate and consent to the study and who have a parent willing to participate.
* Patients with symptoms of minimum three times per week for a duration of two months or greater
* Intact external ear that is free of infection or severe dermatological conditions.
* Stable vital signs for their respective age

Exclusion Criteria:

* Medically complex children or those who take a medication or suffer from an organic disease that can explain symptoms will be excluded from participation.
* Children or parents, who have developmental delay, will be excluded due to difficulties in accurately completing the questionnaires and assessing symptoms.
* History of seizures
* Currently implanted electrical device
* Orthostatic hypotension

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katja Kovacic, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sator-Katzenschlager SM, Wolfler MM, Kozek-Langenecker SA, Sator K, Sator PG, Li B, Heinze G, Sator MO. Auricular electro-acupuncture as an additional perioperative analgesic method during oocyte aspiration in IVF treatment. Hum Reprod. 2006 Aug;21(8):2114-20. doi: 10.1093/humrep/del110. Epub 2006 May 5. PMID 16679325
- [Result] Sator-Katzenschlager SM, Szeles JC, Scharbert G, Michalek-Sauberer A, Kober A, Heinze G, Kozek-Langenecker SA. Electrical stimulation of auricular acupuncture points is more effective than conventional manual auricular acupuncture in chronic cervical pain: a pilot study. Anesth Analg. 2003 Nov;97(5):1469-1473. doi: 10.1213/01.ANE.0000082246.67897.0B. PMID 14570667
- [Result] Asher GN, Jonas DE, Coeytaux RR, Reilly AC, Loh YL, Motsinger-Reif AA, Winham SJ. Auriculotherapy for pain management: a systematic review and meta-analysis of randomized controlled trials. J Altern Complement Med. 2010 Oct;16(10):1097-108. doi: 10.1089/acm.2009.0451. PMID 20954963
- [Result] Busch V, Zeman F, Heckel A, Menne F, Ellrich J, Eichhammer P. The effect of transcutaneous vagus nerve stimulation on pain perception--an experimental study. Brain Stimul. 2013 Mar;6(2):202-9. doi: 10.1016/j.brs.2012.04.006. Epub 2012 May 7. PMID 22621941
- [Result] Kraus T, Kiess O, Hosl K, Terekhin P, Kornhuber J, Forster C. CNS BOLD fMRI effects of sham-controlled transcutaneous electrical nerve stimulation in the left outer auditory canal - a pilot study. Brain Stimul. 2013 Sep;6(5):798-804. doi: 10.1016/j.brs.2013.01.011. Epub 2013 Feb 13. PMID 23453934
- [Result] Sator-Katzenschlager SM, Scharbert G, Kozek-Langenecker SA, Szeles JC, Finster G, Schiesser AW, Heinze G, Kress HG. The short- and long-term benefit in chronic low back pain through adjuvant electrical versus manual auricular acupuncture. Anesth Analg. 2004 May;98(5):1359-64, table of contents. doi: 10.1213/01.ane.0000107941.16173.f7. PMID 15105215
- [Derived] Krasaelap A, Sood MR, Li BUK, Unteutsch R, Yan K, Nugent M, Simpson P, Kovacic K. Efficacy of Auricular Neurostimulation in Adolescents With Irritable Bowel Syndrome in a Randomized, Double-Blind Trial. Clin Gastroenterol Hepatol. 2020 Aug;18(9):1987-1994.e2. doi: 10.1016/j.cgh.2019.10.012. Epub 2019 Oct 14. PMID 31622740
- [Derived] Kovacic K, Hainsworth K, Sood M, Chelimsky G, Unteutsch R, Nugent M, Simpson P, Miranda A. Neurostimulation for abdominal pain-related functional gastrointestinal disorders in adolescents: a randomised, double-blind, sham-controlled trial. Lancet Gastroenterol Hepatol. 2017 Oct;2(10):727-737. doi: 10.1016/S2468-1253(17)30253-4. Epub 2017 Aug 18. PMID 28826627

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects ages 11-18 years, recruited from the outpatient Gastroenterology clinic at the Children's Hospital of Wisconsin between September 2015 and November 2016.
Pre-assignment Details: Subjects were excluded if there were any changes to their current medications or any new medications added during the two weeks prior to study start. Any subject with a new diagnosis of an organic medical condition was also excluded.
Groups:
- Sham Neurostimulator: Inactive auricular neurostimulator treatment x 5 days each week for 4 consecutive weeks
  Sham: Inactive neurostimulator device (without electrical charge), worn for 5 days each week x 4 weeks.
Period: Overall Study
Arm/Group | Neurostimulator | Sham Neurostimulator
Started | 60 | 55
Completed | 57 | 47
Not Completed | 3 | 8
Not completed — Organic disorder diagnosed | 2 | 1
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neurostimulator | Sham Neurostimulator | Total
Number analyzed (Participants) | 57 | 47 | 104
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 15.3 [13.5 to 16.6] | 15.6 [14.7 to 17.2] | 15.3 [13.7 to 16.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 43 | 94
  Male | 6 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 49 | 44 | 93
  Ethnicity: African American | 6 | 2 | 8
  Ethnicity: Hispanic | 1 | 1 | 2
  Ethnicity: Asian | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 47 | 104

OUTCOME MEASURES:

1. Primary Outcome: Pain Frequency-Severity-Duration Scale (PFSD) Score
Description: One-page, 6-item pain measure assessing pain symptoms over the past week. Measures the typical and worst pain intensity, frequency and duration over the past week in units on a scale from 0 to 10 (10 being the worst pain imaginable). Worst pain = primary outcome.
Time Frame: Change from Baseline to Week 4
Population: Modified intent to treat population (all subjects who received minimum one week of therapy and with at least two available data points). Last observation carried forward (LOCF) imputation method.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Neurostimulator | Sham Neurostimulator
Number analyzed (Participants) | 57 | 47
units on a scale | 5.0 [4.0 to 7.0] | 7.0 [5.0 to 9.0]
Statistical Analysis 1: Comparison: Neurostimulator vs Sham Neurostimulator; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 2.15, 95% CI 2-sided [1.37 to 2.93], Standard Error of Mean 0.3947

2. Secondary Outcome: Nausea Profile
Description: Two page, 17-item questionnaire which measures the subjective experience of nausea on a scale from 0 (not at all) to 9 (severely) across three dimensions: 1) somatic distress; 2) gastrointestinal distress and 3) emotional distress. Total score 153.
Time Frame: Change from Baseline to week 4 in Nausea Profile score.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Neurostimulator | Sham Neurostimulator
Number analyzed (Participants) | 57 | 47
units on a scale | 25.5 [11.8 to 43.0] | 20.0 [8.0 to 31.5]

3. Secondary Outcome: State-Trait Anxiety Inventory for Children (STAI-C)
Description: State-Trait Anxiety Inventory for Children (STAI-C). State anxiety measured by 20-item questionnaire assessing anxiety at a particular moment in time on a 3-point rating scale. Raw scores (range 20-60) were converted to normalized T-Scores based on a population of healthy school children (mean=50; standard deviation=10) with higher score indicating worse outcome. Effects of intervention on state anxiety was assessed before (pre) and after (post) therapy.
Time Frame: Change from Baseline (Pre) to 2-3 months after end of therapy (Post)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Neurostimulator | Sham Neurostimulator
Number analyzed (Participants) | 49 | 42
T-score
  State Anxiety Pre | 54.0 [49.0 to 60.5] | 54.0 [46.0 to 56.0]
  State Anxiety Post | 52.0 [46.0 to 58.5] | 54.0 [49.0 to 58.0]

4. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Pediatric Global Health (PGH-7)
Description: A 7-item instrument that measures quality of life in relation to health. Each question has five response options (scored 1-5 units on a scale). A total raw sum score is generated, ranging from lowest score of 7 and highest score of 35 with higher scores indicating better outcome (improved quality of life). The raw score is converted to a standardized T-score (mean=50; standard deviation=10) based on a population of healthy children. T-scores were compared before (Pre) and after (Post) treatment intervention.
Time Frame: Change from Baseline (Pre) to 2-3 months after end of therapy (Post)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Neurostimulator | Sham Neurostimulator
Number analyzed (Participants) | 50 | 43
T-score
  PROMIS Pre | 42.1 [35.6 to 45.7] | 37.2 [34.0 to 43.9]
  PROMIS Post | 42.1 [36.4 to 46.6] | 38.8 [34.0 to 42.1]

5. Secondary Outcome: Functional Disability Inventory (FDI)
Description: 15-item instrument, each question rated on a five-point scale (0="no trouble" to 4="impossible"), indicating how much difficulty subjects have doing common childhood activities because of their physical health. A total score is summed (range 0-60) with higher score indicating worse outcome (greater pain-related disability). Scored were compared before (Pre) and after (Post) treatment intervention.
Time Frame: Change from Baseline (Pre) to 2-3 months after end of therapy (Post)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Neurostimulator | Sham Neurostimulator
Number analyzed (Participants) | 50 | 43
units on a scale
  FDI Pre | 17.0 [7.8 to 27.5] | 17.0 [11.0 to 29.0]
  FDI Post | 11 [6.0 to 22.3] | 17.0 [6.0 to 26.0]

6. Other Pre Specified Outcome: Questionnaire on Pediatric Gastrointestinal Symptoms, Rome III (QPGS-RIII), Reporting the Number of Participants With Specific Diagnoses
Description: Nine-page, validated, parent-report questionnaire that assesses symptoms associated with pediatric functional GI disorders to diagnose the following specific Rome III criteria: Irritable Bowel Syndrome, Functional Dyspepsia, Abdominal Migraine, Functional Abdominal Pain and Functional Abdominal Pain Syndrome. The number of participants with these specific diagnoses at baseline were reported, including overlapping diagnoses.
Time Frame: Baseline only (diagnostic criteria)
Measure: Count of Participants; unit: Participants
Arm/Group | Neurostimulator | Sham Neurostimulator
Number analyzed (Participants) | 57 | 47
Participants
  Irritable Bowel Syndrome | 28 | 23
  Functional Dyspepsia | 12 | 11
  Abdominal Migraine | 16 | 13
  Functional Abdominal Pain | 1 | 0

ADVERSE EVENTS:
Time Frame: 1.5 years (during time of subject participation and through follow-up period)
Description: Information on any adverse events were systematically collected by the research staff at each visit prior to placement of a new neurostimulator and at the follow-up visit.
Arm/Group | Neurostimulator | Sham Neurostimulator
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/47
Other Adverse Events (participants affected / at risk) | 4/57 | 6/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neurostimulator (N=57) | Sham Neurostimulator (N=47)
Ear discomfort (General disorders) | 3 (3) | 3 (3)
Adhesive allergy (Immune system disorders) | 1 (1) | 2 (2) — localized skin irritation
Syncope (Nervous system disorders) | 0 (0) | 1 (1) — triggered by needle phobia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No